CLINICAL TRIAL: NCT06964360
Title: Clinical Trial on Deprescribing Associated With a Psychoeducational Program Using Virtual Reality for Patients With Chronic Pain and Central Sensitization
Acronym: REDOCVR_AC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Badalona Serveis Assistencials (Other)
Responsible Party: Principal Investigator, Jose Ferrer Costa, Medical Researcher and Project Manager, Badalona Serveis Assistencials
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 24/211-ACps
Record Dates: First submitted 2025-05-01; First posted 2025-05-09 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Chronic Pain; Central Sensitisation; Opioid-Related Disorders; Patient Empowerment
Keywords: Virtual Reality; Deprescribing; Primary Health Care; Psychoeducation; Non-Pharmacological Treatment; Emotional Regulation
MeSH Terms: conditions — Chronic Pain; Opioid-Related Disorders; Patient Participation; Emotional Regulation

STUDY DESIGN:
Intervention Model Description: Two groups: REDOCVR intervention vs. standard education control
Masking Description: Not applicable - participants and providers are aware of group assignment due to the nature of the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- REDOCVR Psychoeducational Program (Experimental): Participants receive the full REDOCVR program, a group-based psychoeducational intervention enhanced with immersive virtual reality (VR). The program includes education on pain neuroscience, emotional regulation techniques, physical activation exercises, and VR-based experiential modules. Family physicians provide structured support for supervised tapering of chronic pain medications. The intervention is delivered over 8 weekly sessions of 90 minutes.
  Interventions: Behavioral: REDOCVR Psychoeducational Program
- Control - Standard Education (Active Comparator): Participants receive standard written and audiovisual educational materials related to chronic pain self-management. No virtual reality or group intervention is provided. Participants continue with usual care and may receive general support from their primary care physician, but without structured deprescribing guidance.
  Interventions: Behavioral: Standard Educational Materials

INTERVENTIONS:
Behavioral: REDOCVR Psychoeducational Program — A clinician-guided, group-based psychoeducational program combining pain neuroscience education, emotional regulation techniques, physical activation, and immersive virtual reality experiences. Delivered in eight weekly 90-minute sessions. Includes structured medication tapering support provided by primary care physicians.
  Other Names: Virtual Reality-Enhanced Group Intervention
  Arms: REDOCVR Psychoeducational Program
Behavioral: Standard Educational Materials — Participants receive written and audiovisual materials on chronic pain self-management. Materials are used independently without group sessions or virtual reality. No structured tapering support is provided beyond usual care.
  Other Names: Self-Directed Chronic Pain Education
  Arms: Control - Standard Education

SUMMARY:
This clinical trial evaluates the effectiveness of the REDOCVR program, an interdisciplinary, psychoeducational intervention designed to support deprescribing of chronic pain medications in primary care. REDOCVR integrates group-based education, physical activation, and emotional regulation techniques, enhanced by immersive virtual reality (VR) content that reinforces therapeutic learning and engagement. Rather than functioning as a standalone tool, VR serves as a complementary catalyst within a person-centered, clinician-guided framework. This randomized trial adds a structured medication tapering component and runs in parallel with a complementary pilot study (ClinicalTrials.gov Identifier: NCT06361706), which evaluates the base REDOCVR program without supervised deprescribing. Both protocols are active and jointly contribute to an adaptive, scalable model of chronic pain care in primary care settings. Outcomes include medication use, emotional well-being, anxiety and depression, quality of life, and usability of VR.

DETAILED DESCRIPTION:
This study is part of the broader REDOCVR initiative, a scalable chronic pain management program developed and implemented across primary care centers within Badalona Serveis Assistencials (BSA) in Catalonia, Spain. The REDOCVR program was designed in response to the increasing need for non-pharmacological interventions for chronic pain and integrates psychoeducation, physical activation, and emotional regulation techniques. Immersive virtual reality (VR) is incorporated not as a standalone treatment, but as an enhancing tool to increase engagement, support therapeutic learning, and promote self-management.

This randomized controlled trial represents a complementary arm of the REDOCVR implementation strategy. While the original pilot study (ClinicalTrials.gov Identifier: NCT06361706) focuses on feasibility, usability, and acceptability of the base REDOCVR intervention, the current protocol (24/211-ACps) adds a structured, physician-supervised medication tapering component for patients on chronic pain pharmacotherapy. Both protocols are active and interrelated, reflecting a modular, adaptive implementation model across different primary care sites.

Participants are adults with chronic non-cancer pain, referred during routine clinical visits and screened according to standardized eligibility criteria. The intervention group receives the full REDOCVR program, including immersive VR and deprescribing support, while the control group receives standard educational materials and usual care. Primary and secondary outcomes include change in medication use, emotional well-being (WEMWBS-7), anxiety and depression (HADS), central sensitization (CSI), health-related quality of life (EQ-5D-5L), and usability and satisfaction with the VR platform. Data collection occurs at baseline, post-intervention, and follow-up.

The study follows a hybrid type-2 implementation-effectiveness design and is aligned with ethical and regulatory standards, including approval from the CEIm IDIAPJGol. Findings will contribute to the growing evidence base for interdisciplinary, technology-enhanced models of chronic pain care in real-world primary care settings.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years) diagnosed with chronic non-cancer pain persisting for at least 3 months
* Assigned to one of the participating primary care centers
* Presence of central sensitization symptoms, emotional distress, kinesophobia, or inadequate response to prior treatments
* Capacity to provide informed consent and complete questionnaires

Exclusion Criteria:

* Acute pain conditions (duration <3 months)
* Severe psychiatric or cognitive impairment
* Uncontrolled vertigo, epilepsy, or major visual/auditory impairments
* Conditions contraindicating use of VR equipment
* Inability to attend scheduled sessions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2024-05-06 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Change in daily dose of chronic pain medications | Baseline, immediately post-program (8 weeks), 3-month follow-up
  Reduction in total daily dosage of prescribed medications used for chronic pain (e.g., opioids, benzodiazepines, NSAIDs), converted into standardized dose equivalents.

SECONDARY OUTCOMES:
Change in emotional well-being measured using the 7-item Warwick-Edinburgh Mental Wellbeing Scale (WEMWBS-7) | Baseline, immediately post-program (8-10 weeks)
  A 7-item self-report scale assessing positive mental health, including aspects of optimism, relaxation, and interpersonal relationships.
  Scale Range: 7 to 35 Interpretation: Higher scores indicate better emotional well-being.
Change in anxiety and depression levels measured using the Hospital Anxiety and Depression Scale (HADS), assessing both anxiety and depression subscales. | Baseline, immediately post-program (8-10 weeks)
  A 14-item self-assessment scale with two subscales: HADS-Anxiety (HADS-A) and HADS-Depression (HADS-D), each containing 7 items.
  Scale Range: 0 to 21 per subscale
  Interpretation:
  0-7: Normal 8-10: Borderline abnormal 11-21: Abnormal Higher scores indicate greater levels of anxiety or depression.
Change in central sensitization symptoms measured using the Central Sensitization Inventory (CSI), a self-report tool for sensitization-related symptoms. | Baseline, immediately post-program (8-10 weeks)
  A 25-item self-report questionnaire assessing symptoms related to central sensitization (e.g., widespread pain, sleep disturbance, fatigue).
  Scale Range: 0 to 100 Interpretation: Higher scores indicate more severe symptoms of central sensitization.
  Scores ≥ 40 suggest clinically relevant central sensitization.
Change in health-related quality of life measured using the EuroQol Five-Dimension Five-Level Questionnaire (EQ-5D-5L) | Baseline, immediately post-program (8-10 weeks)
  Each of the five dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) is rated on a 5-point scale (1 = no problems to 5 = extreme problems), describing 3,125 possible health states.
  Two evaluation methods will be used:
  A validated utility index score, derived using a country-specific value set, ranging from less than 0 (worse than death) to 1 (full health).
  A raw sum score of the five dimension levels (range: 5 to 25) will be used for exploratory pre-post comparisons, with acknowledgment that this method is non-validated and should be interpreted cautiously.

CONTACTS AND LOCATIONS:
Locations (4):
- Spain (4):
  - Primary Care Progrès-Raval, Badalona, Barcelona
  - Primary Care Center Apenins-Montigalà, Badalona, Barcelona
  - Primary Care Center Morera-Pomar, Badalona, Barcelona
  - CAP Montgat- Dr Jardi, Montgat, Barcelona

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) that underlie the results reported in this trial will be made available upon reasonable request. This includes anonymized data related to medication use, questionnaire responses, and outcome measures. Data will be shared for research purposes, subject to approval by the study investigators and in compliance with EU GDPR and local data protection regulations. Requests should be directed to the corresponding investigator at Badalona Serveis Assistencials.

REFERENCES:
- See also: Related Pilot Study on ClinicalTrials.gov — https://clinicaltrials.gov/study/NCT06361706